CLINICAL TRIAL: NCT06272006
Title: The Comparison of Different Root Coverage Techniques Using the Anatomical Recession Area Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anatomical recession
Record Dates: First submitted 2024-02-11; First posted 2024-02-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial compares two gingival recession treatments: Coronally Advanced Flap (CAF) with Connective Tissue Graft (CTG) versus Modified Coronally Advanced Tunnel (MCAT) with CTG. Participants are randomized 1:1 to either intervention. Outcomes assessors are blinded to allocation, ensuring unbiased evaluation of the primary outcome, Anatomical Recession Rate (ARR), and secondary clinical outcomes over a 12-month follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study implements single-blind masking where outcomes assessors are unaware of participants' group assignments to minimize bias. While blinding participants and care providers is not feasible due to the nature of surgical interventions, strict protocols ensure assessors remain blinded to treatment allocation throughout the study, enhancing outcome evaluation objectivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronally Positioned Flap (CPF) with Connective Tissue Graft (CTG) (Experimental): Participants in this arm will receive a Coronally Positioned Flap (CPF) surgery combined with a Connective Tissue Graft (CTG). The CPF technique involves surgically repositioning the gum tissue to cover exposed root surfaces, while the CTG procedure involves transplanting connective tissue to the area of gingival recession to encourage regeneration and coverage of exposed roots. This arm aims to evaluate the effectiveness of CPF with CTG in improving gingival recession and periodontal health.
  Interventions: Procedure: Coronally Positioned Flap with Connective Tissue Graft
- Modified Coronally Advanced Tunnel (MCAT) with Connective Tissue Graft (CTG) (Experimental): This arm involves participants receiving the Modified Coronally Advanced Tunnel (MCAT) procedure along with a Connective Tissue Graft (CTG). The MCAT technique is a less invasive approach that creates a tunnel under the gum through which the connective tissue graft is placed without making significant incisions. This method aims to treat gingival recession by encouraging gum regeneration over the exposed roots, with the goal of improving periodontal outcomes and reducing recession.
  Interventions: Procedure: Modified Coronally Advanced Tunnel with Connective Tissue Graft

INTERVENTIONS:
Procedure: Coronally Positioned Flap with Connective Tissue Graft — his intervention involves surgically repositioning the gum tissue over the exposed tooth root and adding a connective tissue graft. The graft is obtained from the patient's palate and placed in the area of gingival recession to promote tissue regeneration and enhance root coverage. The procedure aims to reduce gingival recession and improve periodontal health.
  Arms: Coronally Positioned Flap (CPF) with Connective Tissue Graft (CTG)
Procedure: Modified Coronally Advanced Tunnel with Connective Tissue Graft — This intervention utilizes a minimally invasive technique to create a tunnel beneath the gum tissue, through which a connective tissue graft is placed. The graft, sourced from the patient's palate, is used to encourage the growth of new gum tissue over the exposed root. This method is designed to minimize trauma and promote faster recovery, aiming to improve root coverage and periodontal outcomes.
  Arms: Modified Coronally Advanced Tunnel (MCAT) with Connective Tissue Graft (CTG)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two treatments for gingival recession. The main questions it aims to answer are:

Which treatment method, Coronally Positioned Flap with Connective Tissue Graft or Modified Coronally Advanced Tunnel with connective tissue graft, is more effective in treating gum recession? How does the Anatomical Recession Rate, a new measurement technique, help in evaluating the success of these treatments?

The patients will be treated with coronally advanced flap or modified coronally advanced tunnel + connective tissue graft to see which method is more effective in reducing gum recession, as measured by using anatomical recession rate.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the success of gingival recession treatment methods of coronally advanced flap (CAF) and modified coronally advanced tunnel (MCAT) by using the anatomical ratio rate (ARR). In the parallel-group two-arm randomized clinical study, 40 randomly assigned participants into CAF and MCAT groups will be enrolled. The assessor and investigator will be masked to the interventions that will be applied.

Intervention (CAF): After local anesthesia, the recipient area will be prepared by making a vertical incision from the mesial and/or distal of the last tooth areas where the recession ends, and by applying split-full-split-thickness incisions along with sulcular and subpapillary incisions, thus releasing the flap to facilitate coronal movement. Afterwards, the anatomical papillae will be deepithelised and the recipient area preparation will be completed by applying SRP to the root surfaces. Then, CTG will be harvested from the palatal region by measuring the dimensions of the recession defect. The obtained CTG will be placed on the root surface and sutured to the anatomical papillae with the resorbable sutures. Then, the flap will be sutured to the anatomical papillae with suspended sutures, completely covering the connective tissue graft. Finally, vertical incisions will be sutured to easily coronally position the flap Intervention (MCAT): A split-thickness envelope flap will be created by performing supraperiosteal undermining with tunnel blades and elevators along the facial surface of the papilla. Undermining will be extended to the apical part of the mucogingival line. In order to coronally position the flap, the papillary region will be elevated in full thickness and a supraperiosteal envelope recipient bed will be created. Then, CTG will be obtained according to the size of the recession defect from the palatal region and placed under the tunnel with guide sutures and positioned on the root surfaces, and then the envelope flap will be sutured by pulling it coronally with double cross sutures to completely cover the CTG.

Primary Outcome Measure:

Anatomical Recession Rate (ARR): The primary outcome measure is the Anatomical Recession Rate (ARR), which quantifies the effectiveness of the Coronally Positioned Flap (CPF) with Connective Tissue Graft (CTG) and the Modified Coronally Advanced Tunnel (MCAT) with CTG in covering exposed root surfaces. ARR is calculated by measuring the linear distance between the gingival margin and the cementoenamel junction before and after treatment, with improvements in ARR indicating successful root coverage [Time Frame: 12 months post-treatment].

Secondary Outcome Measures:

Clinical Attachment Level (CAL): This secondary outcome measures the change in the clinical attachment level, indicating the health of the periodontal tissue and its attachment to the tooth root. CAL is a critical parameter for assessing periodontal health and the success of root coverage procedures [Time Frame: Baseline, 3, 6, and 12 months post-treatment].

Gingival Thickness (GT): This outcome assesses the change in gingival thickness, measured in millimeters, post-treatment. Increased gingival thickness is associated with better prognosis and sustainability of the root coverage [Time Frame: Baseline and 12 months post-treatment].

Keratinized Tissue Thickness (KTT): This secondary outcome measures the change in keratinized tissue thickness, indicating the improvement in the quantity of keratinized gum tissue post-treatment. An increase in KTT is considered beneficial for periodontal health and stability, as thicker keratinized tissue can better protect underlying bone and tooth roots from bacterial invasion and mechanical trauma. The thickness will be measured using a periodontal probe or ultrasound device, providing a quantitative assessment of the treatment's effectiveness in enhancing gum tissue resilience [Time Frame: Baseline, 3, 6, and 12 months post-treatment].

Wound healing index (WHI): This outcome will be recorded after surgery using the following criteria: score 1 = uneventful healing with no edema, erythema, suppuration, discomfort, or dehiscence; score 2 = uneventful healing with slight edema, erythema, discomfort, or dehiscence, but no suppuration; and score 3 = poor healing with significant edema, erythema, discomfort, flap dehiscence, or suppuration. [Time Frame: 2 weeks post-treatment].

Tissue appearance: This parameter will be scored according to the consistency, contour, color match, keloid formation degree, and contiguity of the treated sites at T3. Consistency will be rated as firm (1p) or spongy (0p); contour as the presence (2p) or absence (0p) of knife-edged and scalloped GM; color match as excellent (3p), good (2p), adequate (1p), or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); and contiguity as the presence (1p) or absence (0p) of each perceptible incision mark [Time Frame: 6 and 12 months post-treatment].

Aesthetic evaluation: Aesthetics will be evaluated according to the five variables of root coverage esthetic score (RES): GM position, marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC). GM position was scored as 0, 3, or 6, whereas each other variable was scored as 0 or 1 [Time Frame: 6 and 12 months post-treatment].

Dentin hypersensitivity: Hypersensitivity will be recorded using a visual analog scale (VAS) (0 = no pain, 10 = extreme pain) after 3-s air blast applied to the cervical portions of the included sites from a triple syringe [Time Frame: Baseline, 6, and 12 months post-treatment].

Eligibility criteria Minimum Age: 18 Years Maximum Age: 60 Years Sex: All Gender Based: No Accepts Healthy Volunteers: Yes

Inclusion Criteria:

Participants aged 18 to 60 years. Individuals with the gingival recession of Miller Class I, II, or III in at least one tooth in the anterior mandibular or maxillary region.

Participants must have at least 1 mm of keratinized tissue width around the affected tooth/tooth and be in good general health.

Ability to provide informed consent for participation in the study.

Exclusion Criteria:

Individuals with uncontrolled systemic diseases that could impact periodontal healing (e.g., diabetes mellitus, cardiovascular diseases).

Current smokers or those who have quit smoking less than 6 months before the study.

Women who are pregnant or breastfeeding. Participants who have received periodontal or gingival recession treatment in the study area within the last year.

Presence of acute periodontal or dental infections requiring immediate treatment, or extensive caries affecting the study teeth.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 60 years.
* Individuals with the gingival recession of Miller Class I, II, or III in at least one tooth in the anterior mandibular or maxillary region.
* Participants must have at least 1 mm of keratinized tissue width around the affected tooth/tooth and be in good general health.
* Ability to provide informed consent for participation in the study.

Exclusion Criteria:

* Individuals with uncontrolled systemic diseases that could impact periodontal healing (e.g., diabetes mellitus, cardiovascular diseases).
* Current smokers or those who have quit smoking less than 6 months before the study.
* Women who are pregnant or breastfeeding.
* Participants who have received periodontal or gingival recession treatment in the study area within the last year.
* Presence of acute periodontal or dental infections requiring immediate treatment, or extensive caries affecting the study teeth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Anatomical Recession Rate (ARR) | 12 months post-treatment
  The primary outcome measure is the Anatomical Recession Rate (ARR), which quantifies the effectiveness of the Coronally Positioned Flap (CPF) with Connective Tissue Graft (CTG) and the Modified Coronally Advanced Tunnel (MCAT) with CTG in covering exposed root surfaces. ARR is calculated by measuring the linear distance between the gingival margin and the cementoenamel junction before and after treatment, with improvements in ARR indicating successful root coverage.

SECONDARY OUTCOMES:
Clinical Attachment Level (CAL) | Baseline, 3, 6, and 12 months post-treatment
  This secondary outcome measures the change in the clinical attachment level, indicating the health of the periodontal tissue and its attachment to the tooth root. CAL is a critical parameter for assessing periodontal health and the success of root coverage procedures.
Gingival Thickness (GT) | Baseline and 12 months post-treatment
  This outcome assesses the change in gingival thickness, measured in millimeters, post-treatment. Increased gingival thickness is associated with better prognosis and sustainability of the root coverage.
Keratinized Tissue Thickness (KTT) | Baseline, 3, 6, and 12 months post-treatment
  This secondary outcome measures the change in keratinized tissue thickness, indicating the improvement in the quantity of keratinized gum tissue post-treatment. An increase in KTT is considered beneficial for periodontal health and stability, as thicker keratinized tissue can better protect underlying bone and tooth roots from bacterial invasion and mechanical trauma. The thickness will be measured using a periodontal probe or ultrasound device, providing a quantitative assessment of the treatment's effectiveness in enhancing gum tissue resilience.
Wound healing index (WHI) | 2 weeks post-treatment
  This outcome measures the healing by using the following criteria: score 1 = uneventful healing with no edema, erythema, suppuration, discomfort, or dehiscence; score 2 = uneventful healing with slight edema, erythema, discomfort, or dehiscence, but no suppuration; and score 3 = poor healing with significant edema, erythema, discomfort, flap dehiscence, or suppuration
Tissue appearance | 6 and 12 months post-treatment
  This parameter will be scored according to the consistency, contour, color match, keloid formation degree, and contiguity of the treated sites at T3. Consistency will be rated as firm (1p) or spongy (0p); contour as the presence (2p) or absence (0p) of knife-edged and scalloped GM; color match as excellent (3p), good (2p), adequate (1p), or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); and contiguity as the presence (1p) or absence (0p) of each perceptible incision mark
Aesthetic evaluation | 6 and 12 months post-treatment
  Aesthetics will be evaluated according to the five variables of root coverage esthetic score (RES): GM position, marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC). GM position was scored as 0, 3, or 6, whereas each other variable was scored as 0 or 1
Dentin hypersensitivity | Baseline, 6, and 12 months post-treatment
  Hypersensitivity will be recorded using a visual analog scale (VAS) (0 = no pain, 10 = extreme pain) after 3-s air blast applied to the cervical portions of the included sites from a triple syringe

CONTACTS AND LOCATIONS:
Overall Officials: Gencay Keceli, PHD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)